CLINICAL TRIAL: NCT03136341
Title: A Placebo-controlled, Double-blind, Randomized, Cross Over Pilot Study of the Efficacy and Tolerability of Abobotulinum Toxin A (Dysport) as a Treatment for Task-dependent Upper Limb Tremor
Brief Title: A Cross Over Pilot Study of Abobotulinum Toxin A (Dysport) as a Treatment for Task-dependent Upper Limb Tremor
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: David M. Simpson (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor-Investigator, David M. Simpson, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 17-0592
Record Dates: First submitted 2017-04-21; First posted 2017-05-02 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Tremor, Limb
Keywords: Upper Limb; Tremor; task-dependent
MeSH Terms: conditions — Tremor | interventions — abobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive either study drug or placebo at the initial phase and cross over 12 weeks later and receive the alternative treatment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Videos will be randomly provided to an outside assessor to determine benefit as a secondary outcome measure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abobotulinum toxin A (Active Comparator)
  Interventions: Drug: Abobotulinum toxin A
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Abobotulinum toxin A — Dosing will be determined at each study visit based upon muscles involved
  Arms: Abobotulinum toxin A
Other: Placebo — Dosing will be determined at each study visit based upon muscles involved
  Arms: Placebo

SUMMARY:
Task-dependent upper limb tremor is a disorder that frequently impairs patients' function and quality of life. Few studies exist that quantify the improvements in motor performance and disability with botulinum toxin (injections). The study team aims to perform an exploratory pilot trial using toxin Type A (Dysport) in 25 patients with task-dependent upper limb tremor, to refine quantitative measures of performance using blinded video analysis, demonstrate efficacy and tolerability of injections, and provide power calculations for a potential future multi-centered double blinded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with task-dependent essential tremor in upper limb. Tremor is present during at least one of the study functional tasks i. pointing task (touch between nose and a pen held 2 ft. in front. ii. pouring task (cup: pouring water out/in). iii. feeding task (weighted fork from plate on table to mouth). iv. string instrument bowing or holding instrument in static position. v. computer mouse (simple vertical or horizontal movements).
* Patients must be capable of performing informed consent.
* Patients on stable medications for treatment of task-dependent essential tremor for 1 month prior to study entry and maintain them throughout the study.
* Patients previously treated with BoNT of any type must have occurred no sooner than 12 weeks prior to study entry.

Exclusion Criteria:

* Patients with no presence of tremor during study functional tasks.
* Presence of tremor during the functional task is below minimum amplitude required to be considered for injection based upon investigator's clinical judgment.
* Patients with unstable medical conditions or psychiatric conditions.
* Patients with a medical condition that precludes them from receiving BoNT injections.
* Pregnant women, or premenopausal women not willing to use contraceptive measures throughout the duration of the study.
* Lithium, Valproic acid, Amiodarone, typical and atypical neuroleptics. Exposure to other than the listed tremorogenic or potentially tremorogenic drugs is allowed only if, in the opinion of the investigator, this will not interfere with the study drug evaluations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patient's Impression of Change | Week 6
  The principal outcome measure will be patient's impression of change using visual analog scale. Visual Analog Scale (VAS) 100 point scale from 0 (no improvement) to 100 (normal use).
Patient's Impression of Change | Week 18
  The principal outcome measure will be patient's impression of change using visual analog scale. Visual Analog Scale is a 100 point scale from 0 (no improvement) to 100 (normal use).

SECONDARY OUTCOMES:
Physician Global Impression of Change | Week 6
  Physician global impression of change is measured by using a visual analog scale. The CGI using a VAS is rated on a 100-point scale, with the severity of illness scale using a range of responses from 0 (no improvement) through to 100 (normal use).illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).

CONTACTS AND LOCATIONS:
Overall Officials: David M Simpson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jankovic J, Ashoori A. Movement disorders in musicians. Mov Disord. 2008 Oct 30;23(14):1957-65. doi: 10.1002/mds.22255. PMID 18785647
- [Background] Pullman SL, Hristova AH. Musician's dystonia. Neurology. 2005 Jan 25;64(2):186-7. doi: 10.1212/01.WNL.0000157497.08500.c1. No abstract available. PMID 15668411
- [Background] Altenmuller E. Focal dystonia: advances in brain imaging and understanding of fine motor control in musicians. Hand Clin. 2003 Aug;19(3):523-38, xi. doi: 10.1016/s0749-0712(03)00043-x. PMID 12945651
- [Background] Frucht SJ, Fahn S, Greene PE, O'Brien C, Gelb M, Truong DD, Welsh J, Factor S, Ford B. The natural history of embouchure dystonia. Mov Disord. 2001 Sep;16(5):899-906. doi: 10.1002/mds.1167. PMID 11746620
- [Background] Elbert T, Pantev C, Wienbruch C, Rockstroh B, Taub E. Increased cortical representation of the fingers of the left hand in string players. Science. 1995 Oct 13;270(5234):305-7. doi: 10.1126/science.270.5234.305. PMID 7569982
- [Background] Munte TF, Altenmuller E, Jancke L. The musician's brain as a model of neuroplasticity. Nat Rev Neurosci. 2002 Jun;3(6):473-8. doi: 10.1038/nrn843. PMID 12042882
- [Background] Altenmuller E, Jabusch HC. Focal dystonia in musicians: phenomenology, pathophysiology, triggering factors, and treatment. Med Probl Perform Art. 2010 Mar;25(1):3-9. PMID 20795373
- [Background] Schuele S, Jabusch HC, Lederman RJ, Altenmuller E. Botulinum toxin injections in the treatment of musician's dystonia. Neurology. 2005 Jan 25;64(2):341-3. doi: 10.1212/01.WNL.0000149768.36634.92. PMID 15668436
- [Background] Pullman SL, Greene P, Fahn S, Pedersen SF. Approach to the treatment of limb disorders with botulinum toxin A. Experience with 187 patients. Arch Neurol. 1996 Jul;53(7):617-24. doi: 10.1001/archneur.1996.00550070055012. PMID 8929169
- [Background] Carruthers J, Fournier N, Kerscher M, Ruiz-Avila J, Trindade de Almeida AR, Kaeuper G. The convergence of medicine and neurotoxins: a focus on botulinum toxin type A and its application in aesthetic medicine--a global, evidence-based botulinum toxin consensus education initiative: part II: incorporating botulinum toxin into aesthetic clinical practice. Dermatol Surg. 2013 Mar;39(3 Pt 2):510-25. doi: 10.1111/dsu.12148. PMID 23458295
- [Background] Pavicic T, Prager W, Kloppel M, Ravichandran S, Galatoire O. IncobotulinumtoxinA use in aesthetic indications in daily practice: a European multicenter, noninterventional, retrospective study. Clin Cosmet Investig Dermatol. 2015 Mar 5;8:135-42. doi: 10.2147/CCID.S74519. eCollection 2015. PMID 25834463
- [Background] Brin MF, Lyons KE, Doucette J, Adler CH, Caviness JN, Comella CL, Dubinsky RM, Friedman JH, Manyam BV, Matsumoto JY, Pullman SL, Rajput AH, Sethi KD, Tanner C, Koller WC. A randomized, double masked, controlled trial of botulinum toxin type A in essential hand tremor. Neurology. 2001 Jun 12;56(11):1523-8. doi: 10.1212/wnl.56.11.1523. PMID 11402109
- [Background] Louis ED, Barnes L, Wendt KJ, Ford B, Sangiorgio M, Tabbal S, Lewis L, Kaufmann P, Moskowitz C, Comella CL, Goetz CC, Lang AE. A teaching videotape for the assessment of essential tremor. Mov Disord. 2001 Jan;16(1):89-93. doi: 10.1002/1531-8257(200101)16:13.0.co;2-l. PMID 11215599
- [Background] Troster AI, Pahwa R, Fields JA, Tanner CM, Lyons KE. Quality of life in Essential Tremor Questionnaire (QUEST): development and initial validation. Parkinsonism Relat Disord. 2005 Sep;11(6):367-73. doi: 10.1016/j.parkreldis.2005.05.009. PMID 16103000